CLINICAL TRIAL: NCT03015454
Title: A Randomized Controlled Clinical Trial of an Algorithm Driven Sepsis Prediction Biomarker
Brief Title: An Algorithm Driven Sepsis Prediction Biomarker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dascena (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 16-19647
Record Dates: First submitted 2016-12-31; First posted 2017-01-10 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Sepsis; Septic Shock; Severe Sepsis
Keywords: InSight; Dascena
MeSH Terms: conditions — Sepsis; Shock, Septic

ARMS (2):
- With InSight (Experimental): Healthcare provider receives an alert from InSight for patients trending towards severe sepsis. Healthcare provider also receives information from the severe sepsis detector in the UCSF electronic health record.
  Interventions: Other: Severe Sepsis Prediction; Other: Severe Sepsis Detection
- Without InSight (Active Comparator): Healthcare provider does not receive any alerts from InSight. Healthcare provider receives information from the severe sepsis detector in the UCSF electronic health record.
  Interventions: Other: Severe Sepsis Detection

INTERVENTIONS:
Other: Severe Sepsis Prediction — Upon receiving an InSight alert, healthcare provider follows standard practices in assessing possible (severe) sepsis and intervening accordingly.
  Arms: With InSight
Other: Severe Sepsis Detection — Upon receiving information from the severe sepsis detector in the UCSF electronic health record, healthcare provider follows standard practices in assessing possible (severe) sepsis and intervening accordingly.

SUMMARY:
A sepsis early warning predictive algorithm, InSight, has been developed and validated on a large, diverse patient cohort. In this prospective study, the ability of InSight to predict severe sepsis patients is investigated. Specifically, InSight is compared with a well established severe sepsis detector in the UCSF electronic health record (EHR).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the participating units will be eligible.

Exclusion Criteria:

* All patients younger than 18 years of age will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-12; Primary Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Through study completion, an average of 45 days

SECONDARY OUTCOMES:
In-hospital mortality | Through study completion, an average of 45 days

OTHER OUTCOMES:
ICU length of stay | Through study completion, an average of 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Ritankar Das, Principal Investigator — Dascena
Locations (1):
- UCSF Moffit-Long Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Calvert JS, Price DA, Barton CW, Chettipally UK, Das R. Discharge recommendation based on a novel technique of homeostatic analysis. J Am Med Inform Assoc. 2017 Jan;24(1):24-29. doi: 10.1093/jamia/ocw014. Epub 2016 Mar 28. PMID 27026611
- [Background] Calvert J, Desautels T, Chettipally U, Barton C, Hoffman J, Jay M, Mao Q, Mohamadlou H, Das R. High-performance detection and early prediction of septic shock for alcohol-use disorder patients. Ann Med Surg (Lond). 2016 May 10;8:50-5. doi: 10.1016/j.amsu.2016.04.023. eCollection 2016 Jun. PMID 27489621
- [Background] Calvert JS, Price DA, Chettipally UK, Barton CW, Feldman MD, Hoffman JL, Jay M, Das R. A computational approach to early sepsis detection. Comput Biol Med. 2016 Jul 1;74:69-73. doi: 10.1016/j.compbiomed.2016.05.003. Epub 2016 May 12. PMID 27208704
- [Background] Desautels T, Calvert J, Hoffman J, Jay M, Kerem Y, Shieh L, Shimabukuro D, Chettipally U, Feldman MD, Barton C, Wales DJ, Das R. Prediction of Sepsis in the Intensive Care Unit With Minimal Electronic Health Record Data: A Machine Learning Approach. JMIR Med Inform. 2016 Sep 30;4(3):e28. doi: 10.2196/medinform.5909. PMID 27694098
- [Derived] Shimabukuro DW, Barton CW, Feldman MD, Mataraso SJ, Das R. Effect of a machine learning-based severe sepsis prediction algorithm on patient survival and hospital length of stay: a randomised clinical trial. BMJ Open Respir Res. 2017 Nov 9;4(1):e000234. doi: 10.1136/bmjresp-2017-000234. eCollection 2017. PMID 29435343